CLINICAL TRIAL: NCT05094466
Title: A Family-Based Approach to Reducing Obesity Risk Among African American Families
Brief Title: Parent and Family Obesity Intervention in Reducing Obesity Risk in Racial Ethnic Minority Families
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2017-0557; NCI-2021-09374 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2017-0557 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-09-15; First posted 2021-10-26 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Obesity-Related Malignant Neoplasm
MeSH Terms: interventions — Behavior Therapy; Counseling; Early Intervention, Educational; Educational Status; Methods; Interviews as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm I (parent intervention) (Experimental): Parents receive health coaching sessions over 50-60 minutes monthly for 6 months. Parents also receive navigation sessions with a lay LHW monthly for 6 months and church-based peer support monthly for 6 months.
  Interventions: Behavioral: Behavioral Intervention; Other: Counseling; Procedure: Discussion; Other: Educational Intervention; Other: Informational Intervention; Other: Interview
- Arm II (family intervention) (Experimental): Family members receive health coaching sessions over 50-60 minutes monthly for 6 months. Family members also receive navigation sessions with a LHW monthly for 6 months and church-based peer support monthly for 6 months.
  Interventions: Behavioral: Behavioral Intervention; Other: Counseling; Procedure: Discussion; Other: Educational Intervention; Other: Informational Intervention; Other: Interview
- Arm III (delayed comparison) (Active Comparator): Participants receive a handbook that includes core content from the parent and family interventions, but without individual support from coaches, LHWs or the church.
  Interventions: Procedure: Discussion; Other: Educational Intervention; Other: Interview

INTERVENTIONS:
Behavioral: Behavioral Intervention — Receive peer support sessions
  Other Names: Behavior Conditioning Therapy; Behavior Modification; Behavior or Life Style Modifications; Behavior Therapy; Behavioral Interventions; Behavioral Modification; Behavioral Therapy; Behavioral Treatment; Behavioral Treatments
  Arms: Arm I (parent intervention); Arm II (family intervention)
Other: Counseling — Receive health coaching sessions
  Other Names: Counseling Intervention
  Arms: Arm I (parent intervention); Arm II (family intervention)
Procedure: Discussion — Attend focus groups
  Other Names: Discuss
Other: Educational Intervention — Receive handbook
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
Other: Informational Intervention — Receive navigation sessions
  Arms: Arm I (parent intervention); Arm II (family intervention)
Other: Interview — Participate in interview

SUMMARY:
This clinical trial compares the effects of parent/caregiver-focused programs to family-focused programs in reducing obesity risk in racial ethnic minority families. Obesity tends to run in families, thus family-based interventions have been strongly recommended. Parent and family obesity programs may reduce obesity risk and ultimately reduce the risk of obesity-related cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Establish the feasibility and acceptability of the Parent and Family obesity interventions.

SECONDARY OBJECTIVES:

I. Explore congregational and community interest in obesity and obesity related behaviors in racial ethnic minorities.

II. Explore the preliminary impact of the Parent and Family interventions on behavioral, social and environmental outcomes in parent/child dyads. III. Explore potential mediators (self-efficacy, perceived stress, depressive symptoms) and moderators (sex of dyads, family history of lifestyle changes, and church attendance).

OUTLINE: Churches are randomized to 1 of 3 arms.

ARM I (PARENT INTERVENTION): Parents receive health coaching sessions over 50-60 minutes monthly for 6 months. Parents also receive navigation sessions with a lay health worker (LHW) monthly for 6 months and church-based peer support monthly for 6 months.

ARM II (FAMILY INTERVENTION): Family members receive health coaching sessions over 50-60 minutes monthly for 6 months. Family members also receive navigation sessions with a LHW monthly for 6 months and church-based peer support monthly for 6 months.

ARM III (DELAYED COMPARISON): Participants receive a handbook that includes core content from the parent and family interventions, but without individual support from coaches, LHWs or the church.

ELIGIBILITY:
Inclusion Criteria:

* ELIGIBLE IN-DEPTH INTERVIEW PARTICIPANTS: Any church leader, such as pastors, minister, church secretary, health ministry leader, youth leader, deacons, ministry leader, director
* PARENT-CHILD DYADS: Be parent/caregiver (legal parent or custodial grandparent; male or female) and child willing to participate
* PARENT-CHILD DYADS: Live together in the same household
* PARENTS/CAREGIVERS: Self-identify as a racial ethnic minority (i.e., black or African American or Hispanic)
* PARENTS/CAREGIVERS: Parent or caregiver age 18 through 65 years old
* PARENTS/CAREGIVERS: Are obese (body mass index [BMI] >= 30)
* PARENTS/CAREGIVERS: Are not currently participating in a physical activity (PA), diet, or weight management program
* PARENTS/CAREGIVERS: Enroll with a child aged 10-16 years
* PARENTS/CAREGIVERS: Have a valid home address, telephone number, and internet access
* PARENTS/CAREGIVERS: Are able to speak, read, and write in English
* CHILDREN: They are aged between 10-16 years

Exclusion Criteria:

* PARENTS/CAREGIVERS: They are currently pregnant or thinking about becoming pregnant during study period
* PARENTS/CAREGIVERS: They present any contraindications for exercise based on responses to the PA Readiness Questionnaire
* PARENTS/CAREGIVERS: Principal investigator (PI) determines that parent/caregiver is unsuitable for the study for reasons not otherwise stated in the protocol

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-07-16 (Actual); Primary Completion 2027-02-02 (Estimated); Study Completion 2027-02-02 (Estimated)

PRIMARY OUTCOMES:
The correlation between the feasibility of the Parent and Family obesity interventions. | Up to 4 years
The correlation between the acceptability of the Parent and Family obesity interventions. | Up to 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Lorna McNeill, PhD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org